CLINICAL TRIAL: NCT01908270
Title: Randomized Controlled Trial of Yoga for Menopausal Symptoms in Women With Breast Cancer
Brief Title: Effects of Yoga on Menopausal Symptoms in Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research Fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-5421-BO
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Menopause; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (Experimental): Yoga intervention 12 weeks, weekly 90-minute intervention Yoga postures, breathing, relaxation, and meditation
  Interventions: Behavioral: Yoga; Other: Usual care
- Usual care (Other): Patients continue usual care by their practitioner
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Yoga
  Arms: Yoga
Other: Usual care

SUMMARY:
Women with breast cancer and breast cancer survivors are often bothered by menopausal symptoms to a special degree. Treatment options for those symptoms are currently limited as hormone replacement therapy is often prohibited. Yoga has been shown to reduce menopausal symptoms as well as symptoms associated with breast cancer. Therefore, this study aims to investigate whether a 12-week yoga intervention can reduce menopausal symptoms in women with breast cancer and breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer (Stage I-III)
* After completion of surgical therapy
* After completion of adjuvant radiotherapy and chemotherapy
* Score of 5 or greater on the Menopausal Rating Scale
* Physical and cognitive capacity to participate in the yoga intervention
* Willingness to participate in 10 or more of the 12 yoga interventions
* signed informed consent

Exclusion Criteria:

* Regular yoga practice in the past 12 months
* Planned surgery in the study period
* Diagnosed and medically treated psychosis
* Hormone replacement therapy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Menopausal symptoms | Week 12
  Menopause Rating Scale

SECONDARY OUTCOMES:
Health-related quality of life (disease-specific) | Week 12
  Functional Assessment of Cancer Therapy - Breast
Fatigue | Week 12
  Functional Assessment of Chronic Illness Therapy - Fatigue
Anxiety | Week 12
  Hospital Anxiety and Depression Scale
Depression | Week 12
  Hospital Anxiety and Depression Scale
Menopausal symptoms | Week 24
  Menopause Rating Scale
Health-related quality of life (disease-specific) | Week 24
  Functional Assessment of Cancer Therapy - Breast
Fatigue | Week 24
  Functional Assessment of Chronic Illness Therapy - Fatigue
Anxiety | Week 24
  Hospital Anxiety and Depression Scale
Depression | Week 24
  Hospital Anxiety and Depression Scale
Adverse events | Week 12
Adverse events | Week 24

OTHER OUTCOMES:
Appraisal of body | Week 12
  Fragebogen zur Beurteilung des Körpers (Questionnaire for the assessment of body)
Appraisal of body | Week 24
  Fragebogen zur Beurteilung des Körpers (Questionnaire for the assessment of body)
Body awareness | Week 12
  Body Awareness Questionnaire
Body awareness | Week 24
  Body Awareness Questionnaire
Self-esteem | Week 12
  Self-esteem scale
Self-esteem | Week 24
  Self-esteem scale
Adherence | Week 12
  Course adherence and daily home practice
Adherence | Week 24
  Daily home practice

CONTACTS AND LOCATIONS:
Overall Officials: Holger Cramer, PhD, Principal Investigator — Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Faculty of Medicine, University of Duisburg-Essen, Essen, Germany